CLINICAL TRIAL: NCT07227610
Title: Brain Metastases in Greater Size - Hypofractionated Options Trial (BIGSHOT)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104122
Record Dates: First submitted 2025-11-10; First posted 2025-11-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Brain Metastases; Cancer (With CNS Involvement)
Keywords: Cancer; Brain
MeSH Terms: conditions — Brain Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Staged Stereotactic Radiosurgery (SSRS) (Experimental): Patient will be scheduled for treatment with SSRS within one week of randomization. The large brain metastasis (or metastases) will be treated to a dose of 24-30 Gy in two fractions. Interval between the two fractions will be 30 days (+/- 10 days). MRI brain for planning purposes will be obtained either on the day of each treatment, or within 7 days prior to each treatment. Individual dosing for each fraction will be determined by the treating radiation oncologist, but total dose must equal 24-30 Gy. Any additional smaller metastases will be treated in a single fraction concurrently. Fixation for treatment will be either in a surgical headframe or mask.
  Interventions: Radiation: Staged Stereotactic Radiosurgery (SSRS)
- Fractionated Stereotactic Radiotherapy (FSRT) (Experimental): Patient will be scheduled for treatment with FSRT within one week of randomization. FSRT will be performed with mask fixation. Fractionation will be 27 Gy in 3 daily fractions. The 3 daily fractions must be completed over a period of 3-5 days. MRI for planning purposes must be completed within 7 days prior to delivery of first fraction. Any additional smaller metastases will be treated in a single fraction concurrently.
  Interventions: Radiation: Fractionated Stereotactic Radiotherapy (FSRT)

INTERVENTIONS:
Radiation: Staged Stereotactic Radiosurgery (SSRS) — The large brain metastasis (or metastases) will be treated to a dose of 24-30 Gy in two fractions. Interval between the two fractions will be 30 days (+/- 10 days). Individual dosing for each fraction will be determined by the treating radiation oncologist, but total dose must equal 24-30 Gy.
  Arms: Staged Stereotactic Radiosurgery (SSRS)
Radiation: Fractionated Stereotactic Radiotherapy (FSRT) — Fractionation will be 27 Gy in 3 daily fractions. The 3 daily fractions must be completed over a period of 3-5 days.
  Arms: Fractionated Stereotactic Radiotherapy (FSRT)

SUMMARY:
This is a randomized, phase II trial comparing staged stereotactic radiosurgery (SSRS) versus fractionated stereotactic radiotherapy (FSRT) in patients with large brain metastases (≥2 cm and ≤5 cm). The study aims to evaluate efficacy, safety, and tumor response between these two standard-of-care radiation approaches.

DETAILED DESCRIPTION:
Brain metastases are an increasingly common diagnosis, as cancer patients continue to live longer due to advances in systemic therapy. Up to 26% of patients with metastatic cancer will develop metastatic disease to the brain (Nayak 2012), most commonly in lung cancer, as well as melanoma, breast, and renal cell cancer (Singh 2020). Historically, brain metastases were treated with whole brain radiation therapy (WBRT). However, increasing evidence over the past 10-15 years, as well as technological advances, have created a shift in treatment toward stereotactic radiosurgery (SRS), which is a focused treatment targeting only the visible tumors. SRS has multiple advantages over WBRT. Most importantly, focused treatment with SRS provides significantly lower risk of neurocognitive toxicity compared with WBRT, with no difference in overall survival (Chang 2009, Brown 2016, Aoyama 2006). SRS is also more convenient, delivered in 1 to 3 treatments, as opposed to 2 weeks of therapy with WBRT. For these reasons, SRS is now the preferred option for patients with limited brain metastases, recognized in both the NCCN guidelines and ASTRO guidelines (Gondi 2022).

For intact metastases less than 2 cm, local control with SRS alone is excellent (Redmond 2021). However, for larger tumors, achieving long term local control with radiation is more difficult. Tumor dosing is based on risk of toxicity (specifically, radiation necrosis), and therefore for larger tumors, the dose is decreased (RTOG 90-05, Johannwerner 2023). This results in suboptimal control for tumors >2 cm. For single fraction SRS, local control is estimated around 70%, and for fractionated SRS (3-5 fractions), around 80% (Redmond 2021).

There are two common approaches for treating large intact brain metastases with radiosurgery alone. Fractionated SRS involves treating the tumor in 3-5 separate daily treatments. This allows for normal tissue recovery in between, and therefore may decrease the risk of toxicity (Minitti 2015). Staged SRS involves treating the tumor in two sessions, spaced apart by 3-6 weeks. This allows delivery of a lower dose for the first fraction (to minimize toxicity), and the second fraction can be dose escalated depending on interval tumor response. A recent meta-analysis compared SSRS to FSRT, and found no difference in local control, but a lower rate of re-treatment in the SSRS group (Harikar 2023). Radiation necrosis rate was 3.7% in the SSRS group and 6.4% in the FSRT group. The authors of this study concluded that randomized controlled trials examining the two options would be useful. A retrospective study conducted a propensity score-matched analysis of SSRS vs FSRT. This study showed comparable rates of local failure (15% at 6 months, and 25% at one year in both groups), as well as comparable rates of radiation necrosis (2.2% in SSRS vs 6.4% in FSRT) (Noda 2023).

In theory, treatment with SSRS would allow for a higher biological equivalent dose (BED) to the target lesion, while maintaining low toxicity rate, as time between fractions allows for normal tissue recovery. Retrospective data suggests that a BED10 > 50 predicts for better one year local control in hypofractionated SRS (Remick 2020). BED10 for 9 Gy x3 is 51.3Gy, with an EQD2 a/b 2 of 74.25. In comparison, 15 Gy x2 results in a BED10 of 75Gy, with EQD2 a/b 2 of 127.5. Allowing 3-6 weeks of recovery time in between the two fractions should theoretically allow for tissue recovery and mitigate the risk of higher normal tissue EQD2. Additionally, while data for 3 fraction FSRT is encouraging for larger tumors (2-5 cm), the local control for tumors on the larger end of this spectrum (>3 cm) may not be as good. Specifically, in one of the largest retrospective studies of 3 fraction FSRT for metastases >2cm, the overall local control was 91% at 1 year; however, the local control for lesions 3 cm or larger was only 73% (Minniti 2015).

Although there is encouraging retrospective data supporting the use of both SSRS and FSRT, there are no studies directly comparing the two approaches in a prospective fashion. Therefore, randomized data is needed to provide guidance on the best approach in this challenging patient population.

This study will compare two approaches for treating large brain metastases (2-5 cm): staged stereotactic radiosurgery (SSRS) and fractionated stereotactic radiotherapy (FSRT). These are both considered standard treatments and both used as standard of care for patients with large brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or a legally authorized representative must be able and willing to provide study-specific informed consent prior to study entry.
2. Patient must be willing to comply with all study procedures and available for the duration of the study
3. Male or female, aged ≥ 18 years
4. Karnofsky Performance Status (KPS) ≥ 60 within 7 days prior to registration
5. Radiographic confirmation of brain metastasis measuring ≥2 cm and ≤ 5 cm in maximum diameter

   1. Multiple metastases are allowed. Additional metastases will be treated with single fraction SRS as per standard of care. Up to 10 additional smaller metastases are allowed on protocol. All additional smaller metastases must be less than 2 cm.
   2. If a patient has more than one large metastasis (measuring between 2 and 5 cm as above), up to two can be treated on study protocol
   3. All tumors must be ≥ 5mm from the optic chiasm and optic nerves.
6. Known active or history of invasive non-CNS primary cancer based on documented pathologic diagnosis within the past 3 years
7. Patient is able to medically tolerate SRS
8. Patient is neurologically stable (immediate surgery not necessary or not recommended)
9. A negative urine or serum pregnancy test (in persons of childbearing potential) within 7 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal.
10. Participants who are sexually active must agree to use medically acceptable forms of contraception during treatment on this study to prevent pregnancy.

Exclusion Criteria:

1. Prior cranial radiotherapy, including whole brain radiotherapy (WBRT), or SRS in the area of the large metastasis to be treated on study.
2. Evidence of leptomeningeal disease (LMD) Note: For the purposes of exclusion, LMD is a clinical diagnosis, defined as positive CSF cytology and/or unequivocal radiologic or clinical evidence of leptomeningeal involvement. Patients with leptomeningeal symptoms in the setting of leptomeningeal enhancement by imaging (MRI) would be considered to have LMD even in the absence of positive CSF cytology. In contrast, an asymptomatic or minimally symptomatic patient with mild or nonspecific leptomeningeal enhancement (MRI) would not be considered to have LMD. In such cases, CSF sampling is not required to formally exclude LMD, but can be performed at the investigator's discretion based on level of clinical suspicion.
3. Inability to undergo MRI with contrast
4. Planned administration of systemic therapy (chemotherapy or immunotherapy) within 3 days prior to, the day of, or 3 days after completion of SRS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2029-02-03 (Estimated); Study Completion 2030-02-03 (Estimated)

PRIMARY OUTCOMES:
Time to Composite unfavorable outcome (CUO) by (1) lack of local control (disease progression for any lesion treated on study); (2) the need for further intervention to the treated tumor; (3) radiation necrosis. | Up to 36 months.
  For lesions > 5 mm: Disease progression is defined as at least a 50% increase in the product of the two longest diameters of the target lesion, compared to the smallest product measured for that lesion.
  For lesions ≤ 5mm on the baseline scan, disease progression is defined as at least a 100% increase in the product of the two longest diameters of the target lesion, compared to the smallest product measured for the same lesion.
  * Radiation necrosis is defined by: pathologic diagnosis after resection or biopsy; OR initiation of steroids, and follow up MRI scan shows decrease in edema and stability of contrast of enhancing lesion that was concerning for radiation necrosis.
  * Radiation necrosis is NOT counted as disease progression.
  * Additional interventions include surgical resection, LITT (laser interstitial thermal therapy), or re-irradiation to the target lesion.

SECONDARY OUTCOMES:
Compare the safety profile by radiation toxicity | Up to 36 months
  Radiation toxicity defined as need for prolonged steroids (>2 weeks) due to symptoms related to the treated tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Rivers, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) may be shared with qualified researchers upon request after the primary endpoint is completed. Requests should be directed to the Medical University of South Carolina.
Time Frame: After completion of the primary endpoint.
Access Criteria: Requests will be reviewed and approved by the study sponsor. Data will be shared in accordance with institutional and NIH policies.